CLINICAL TRIAL: NCT07232563
Title: Exploratory Study of Intranasal Administration of Small Extracellular Vesicles Derived From Human Umbilical Cord Mesenchymal Stem Cells hUC-MSC-sEV-001 in the Treatment of Ischemic Stroke Patients
Brief Title: Exploratory Study of Intranasal Administration of Human Umbilical Cord Mesenchymal Stem Cell-Derived Extracellular Vesicles for the Treatment of Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-343-04
Record Dates: First submitted 2025-09-21; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; stem cell; Extracellular Vesicles
MeSH Terms: conditions — Ischemic Stroke | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal Administration of hUC-MSC-sEV-001 Therapy (Experimental): Intranasal Administration of Human Umbilical Cord Mesenchymal Stem Cell-Derived Small Extracellular Vesicles (hUC-MSC-sEV-001) Therapy
  Interventions: Biological: Intranasal Administration of Human Umbilical Cord Mesenchymal Stem Cell-Derived Small Extracellular Vesicles (hUC-MSC-sEV-001) Therapy

INTERVENTIONS:
Biological: Intranasal Administration of Human Umbilical Cord Mesenchymal Stem Cell-Derived Small Extracellular Vesicles (hUC-MSC-sEV-001) Therapy — Experimental drug: hUC-MSC-SEV-001 nasal drops derived from small extracellular vesicles of human umbilical cord mesenchymal stem cells Treatment plan: On the basis of conventional treatment, hUC-MSC-SEV-001 nasal drops will be administered: hUC-MSC-SEV-001 will be administered via nasal drip for a total of 4 times, with a dosage of 1 × 10 * 11articles per dose. The patient will receive one dose on the day of enrollment, and another dose of hUC-MSC-SEV-001 will be administered on the 2nd, 3rd, and 4th days after enrollment.

SUMMARY:
Evaluation of the Safety and Preliminary Efficacy of Intranasal Administration of Human Umbilical Cord Mesenchymal Stem Cell-Derived Small Extracellular Vesicles (hUC-MSC-sEV-001) in Patients for Ischemic Stroke

DETAILED DESCRIPTION:
Based on adhering to the GCP principles of national clinical trial research and the standardized processes of CROs, this study aims to evaluate the safety and preliminary efficacy of hUC-MSC-sEV-001 in treating ischemic stroke by recruiting a small sample population. Additionally, the study will seek to determine an appropriate dosage, laying the foundation for subsequent research.

ELIGIBILITY:
Inclusion criteria:

* Ischemic Stroke
* Age 18-70 years, no gender restriction
* Confirmed anterior circulation occlusion by CTA or MR angiography (MRA)
* Pre-stroke mRS score of 0-1
* Post-stroke ASPECTS score >= 6
* Pre-enrollment NIHSS score>= 6
* Within 24 hours to 14 days of stroke onset
* Patients who have not received thrombolysis or endovascular treatment
* No significant liver or kidney dysfunction: ALT and AST<= 2.5 times the upper limit of normal, serum creatinine and blood urea nitrogen <= 1.25 times the upper limit of normal
* No significant cardiac dysfunction
* The subject or legal representative can sign the informed consent form and comply with the requirements of the study for administration and follow-up.

Exclusion criteria:

* Intracranial hemorrhagic conditions observed on cranial CT: hemorrhagic stroke, epidural hematoma, subdural hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, or hemorrhagic transformation, etc.
* Known severe allergy to contrast agents (excluding mild rash-type allergies)
* Known bleeding tendencies (including but not limited to): platelet count < 100×10^9/L; received heparin treatment within 48 hours with aPTT >= 35s; currently taking warfarin with INR > 1.7
* Patients with brain tumors, or a history of epilepsy and severe head trauma
* Patients with other systemic malignancies
* Patients with other serious systemic diseases such as immunodeficiency, coagulation disorders, etc.
* Patients with Alzheimer's disease, Parkinson's disease, or other neurodegenerative diseases that prevent them from completing follow-up
* Patients with severe local infection, systemic infection, immunodeficiency, or those currently taking immunosuppressants
* Patients who are positive for hepatitis B surface antigen or currently suffering from other infectious diseases
* Patients who have allergic reactions to the drug used in this study or similar drugs
* Patients with known allergic constitution
* Patients with nasal structural abnormalities or lesions
* Patients with cerebrospinal fluid rhinorrhea
* Patients who have participated in other clinical trials within the past 3 months
* Unwilling or unable to comply with the procedures specified in the protocol
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling or unable to use appropriate contraceptive measures
* Patients clearly lacking the compliance to complete the clinical trial, such as those suffering from uncontrolled mental illness
* Other situations deemed unsuitable for enrollment by the researchers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-07 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) Related to hUC-MSC-sEV-001 | Day 14 (+-2) post-enrollment
  Dose-Limiting Toxicity (DLT) Related to hUC-MSC-sEV-001 Includes:
  1. Grade 3-4 severe adverse events occurring on day 14 (+-2), graded according to Common Terminology Criteria for Adverse Events （CTCAE） V5.0;
  2. NIHSS score increase of ≥4 from baseline on day 14 (+-2); NIHSS score assessed by a professional rehabilitation physician;
  3. Symptomatic intracranial hemorrhage occurring on day 14 (+-2); detected via CT scan and patient symptom presentation.

SECONDARY OUTCOMES:
Serious adverse events related to the investigational drug within 90 (+-7) days | At baseline, Day 7 (+-1), Day 14 (+-2), and Day 90 (+-7)post-enrollment
  The occurrence of serious adverse events related to the investigational drug will be assessed according to CTCAE v5.0, based on monitoring of the patient's vital signs (pulse, blood pressure, respiration, and body temperature), as well as laboratory tests including complete blood count, urinalysis, liver and kidney function, glucose and lipid metabolism, coagulation profile, serum electrolytes, tumor markers, and electrocardiogram.
Distribution of Modified Rankin Scale (mRS) Scores within 90 (+-7) days | baseline, Day 7 (+-1), Day 14 (+-2), and Day 90 (+-7)post-enrollment
  Measured using the Modified Rankin Scale (mRS) scale. The mRS ranges from 0 to 6, with higher numbers indicating greater disability.
Barthel Index within 90 (±7) days | baseline, Day 7 (+-1), Day 14 (+-2), and Day 90 (+-7)post-enrollment
  Measured using the Barthel Index. The total score of the Barthel Index ranges from 0 to 100 points. A higher Barthel Index score indicates a better (more positive) outcome, while a lower score indicates a poorer (more challenging) outcome.
Five-level, five-dimensional EuroQol (EQ-5D-5L) | baseline, Day 7 (+-1), Day 14 (+-2), and Day 90 (+-7)post-enrollment
  Measured using the Five-level, five-dimensional EuroQol (EQ-5D-5L). It has two main scores with distinct ranges. The Index Score (Utility Score) comes from mapping responses on 5 health dimensions to a standardized scale. Its minimum is typically -0.594 to -0.101 (varies by region; negatives mean health worse than death for some), and maximum is 1.0 (full health, no limitations). The Visual Analog Scale (VAS) Score is a subjective self-rating on a 100mm vertical line, with 0 ("Worst imaginable health") as minimum and 100 ("Best imaginable health") as maximum. For both scores, higher means better HRQoL.
Proportion of Modified Rankin Scale (mRS) Scores of 0-2 within 90 (+-7) days | baseline, Day 7 (+-1), Day 14 (+-2), and Day 90 (+-7)post-enrollment
  Measured using the mRS scale
All-cause mortality at 90 (+-7) days | Day 90 (+-7)post-enrollment
  Contact the patient or their family to confirm survival status
Changes in infarct volume at 14 (+-2) days compared to baseline | baseline, Day 14 (+-2) post-enrollment
  Using CTA、 CTP and MRI to measure changes in infarct volume in patients
Change from Baseline in National Institutes of Health Stroke Scale (NIHSS) Score | baseline, Day 7 (+-1) and Day 14 (+-2)post-enrollment
  Measured using the National Institutes of Health Stroke Scale (NIHSS). Its total score range spans from a minimum of 0 points (indicating no detectable neurological deficits, suggesting minimal or no stroke-related impairment) to a maximum of 42 points (representing severe, widespread neurological dysfunction, often associated with profound stroke-related disability); regarding the scoring standard, a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- 253 Gongye Blvd Middle, Guangzhou, Guangdong, China 510280, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data from this trial will be shared through the public data repository"ResMan" after the study results are published. The dataset includes all raw data, processed data, and statistical analysis codes. Data will be anonymized to ensure participant privacy. The data can be accessed via the following link: [www.medresman.org.cn]. For any inquiries, please contact the corresponding author: [zrah@163.com].
Supporting Information: SAP, CSR, Analytic Code
Time Frame: The data from this trial will be shared through the public data repository"ResMan" after the study results are published.

DOCUMENTS (2):
  • Study Protocol (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT07232563/Prot_000.pdf
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT07232563/ICF_001.pdf